CLINICAL TRIAL: NCT03814044
Title: PMCF Study on PEEK Suture Anchors for Hip Indications
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018.14.SMD.PEEK.RET.HIP
Record Dates: First submitted 2018-10-24; First posted 2019-01-23 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-09

CONDITIONS: Soft Tissue to Bone Fixation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PEEK Suture Anchors — Subjects who have undergone hip joint repair using PEEK Suture Anchors:
  BIORAPTOR™ Knotless Suture Anchor and SpeedLock Hip Suture Anchor

SUMMARY:
Post-market clinical follow-up (PMCF) on the PEEK Suture Anchors in the hip.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have undergone hip joint repair using the study devices.
2. Subjects aged 18 years and older at the time of surgery.
3. Subjects who had a visit to their provider between 3 and 15 months postoperative.

Exclusion Criteria:

1. Subjects who are < 12 months post-operative.
2. Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 30 days prior to surgery
3. Subject had off-label use of the PEEK suture anchor during surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone hip joint repair using PEEK Suture Anchors:
  * BIORAPTOR Knotless Suture Anchors
  * SpeedLock Hip
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Horner, Study Chair — Smith & Nephew, Inc.
Locations (4):
- United States (4):
  - DMOS Orthopedic Centers, West Des Moines, Iowa
  - Center for Advanced Orthopedic and Sports Medicine, Auburn Hills, Michigan
  - Community Hospital - Oklahoma City, Oklahoma City, Oklahoma
  - Southwest Orthopaedic Reconstructive Specialists, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 149 participants were enrolled in the study and 150 joints were observed.
Units Other Than Participants: joints
Groups:
- Polyetheretherketone (PEEK) Hip Suture Anchors: Participants who have received PEEK Suture Anchors in the hip which included:
  BIORAPTOR™ Knotless Suture Anchor and SpeedLock Hip Suture Anchor
Period: Overall Study
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Started | 149; 150 joints
BIORAPTOR™ Knotless Suture Anchor | 58; 58 joints
SpeedLock Hip Suture Anchor | 93; 94 joints
Completed | 148; 149 joints
Not Completed | 1; 1 joints
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study who had previously undergone extremity repair using PEEK suture anchors (i.e., retrospective data). The type(s) of PEEK anchor used during surgery was surgeon decision on a case by case basis. Multiple anchor types could be used in one surgery if required. Two participants had multiple devices implanted. Participants with bilateral surgeries had both surgeries recorded independently. Device data analyzed individually dependent on unique suture anchor implanted.
Units Other Than Participants: joints
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Number analyzed (Participants) | 149
Number analyzed (joints) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (11.9)
Sex: Female, Male [Count of Units; unit: joints]
  Female | 105
  Male | 45
Ethnicity (NIH/OMB) [Count of Units; unit: joints]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 52
Race/Ethnicity, Customized [Count of Units; unit: joints]
  American Indian or Alaska Native: No | 149
  American Indian or Alaska Native: Yes | 1
  Asian: No | 150
  Asian: Yes | 0
  Black or African American: No | 147
  Black or African American: Yes | 3
  Native Hawaiian or Other Pacific Islander: No | 150
  Native Hawaiian or Other Pacific Islander: Yes | 0
  White: No | 6
  White: Yes | 144
  Other: No | 147
  Other: Yes | 3
Location of Device Implantation [Count of Participants; unit: Participants]
  Left Hip | 71
  Right Hip | 77
  Bilaterally | 1
Duration of Surgery (min) [Mean (Standard Deviation); unit: minutes] — Population: Data only available for 20 participants due to the retrospective nature of the study.
  minutes
    number analyzed (Participants) | 20
    (all) | 87.4 (11.9)
Intervention [Count of Units; unit: joints]
  Arthroscopic | 150
  Open | 0
  Unknown | 0
Duration of time from injury to surgery (days) [Mean (Standard Deviation); unit: days] — Population: Data only available for 86 participants due to the retrospective nature of the study.
  days
    number analyzed (Participants) | 86
    (all) | 905.6 (823.1)
Any Medical History [Count of Units; unit: joints]
  Yes | 95
  No | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success of the Study Devices in the Hip Over a Time Period of 6 Months After Intervention
Description: Clinical success was defined as hip repairs without signs of device failure and/or re-intervention as assessed by the surgeon (Yes/No). Specifically, clinical success was achieved with "Yes" responses on the following 3 main criteria:
  * no inflammatory or allergic response
  * no device-related adverse event (AE)
  * no device deficiencies (DDs) leading to revision surgery (reintervention) on the index hip
Time Frame: 6 months
Population: Participants analyzed for each row indicate those with available retrospective data for the time frame & outcome specified. 2 participants implanted with multiple Suture Anchors (devices). Data analyzed independently based on device implanted (i.e., participants with multiple devices analyzed by unique suture anchor). Anchors shown by rows/categories as the same procedure occurred on the same joint. Overall number of participants analyzed shows combined total of distinct participants assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Number analyzed (Participants) | 149
Participants
  BIORAPTOR™ Knotless Suture Anchor: number analyzed (Participants) | 58
  BIORAPTOR™ Knotless Suture Anchor: Yes | 58
  BIORAPTOR™ Knotless Suture Anchor: No | 0
  SpeedLock Hip Suture Anchor: number analyzed (Participants) | 93
  SpeedLock Hip Suture Anchor: Yes | 93
  SpeedLock Hip Suture Anchor: No | 0

2. Secondary Outcome: Number of Participants With Clinical Success of the Study Devices in the Hip Over a Time Period of 12 Months After Intervention
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Number analyzed (Participants) | 64
Participants
  BIORAPTOR™ Knotless Suture Anchor: number analyzed (Participants) | 42
  BIORAPTOR™ Knotless Suture Anchor: Yes | 42
  BIORAPTOR™ Knotless Suture Anchor: No | 0
  SpeedLock Hip Suture Anchor: number analyzed (Participants) | 24
  SpeedLock Hip Suture Anchor: Yes | 24
  SpeedLock Hip Suture Anchor: No | 0

3. Secondary Outcome: Visual Analog Scale (VAS) - Pain
Description: The VAS pain score is presented on a scale ranging from 0 to 10. A score of 0 represents no pain and a score of 10 indicates extreme/unbearable pain. The VAS rating was recorded retrospectively, per standard of care at 6 and 12 months post-surgery.
Time Frame: 6 and 12 months
Population: No data were collected at 6 months or 12 months for VAS pain score due to the retrospective nature of the study.
Groups:
- Polyetheretherketone (PEEK) Hip Suture Anchors: Participants who have received PEEK Suture Anchors in the hip which included:
  BIORAPTOR™ Knotless Suture Anchor SpeedLock Hip Suture Anchor
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Number analyzed (Participants) | 0

4. Secondary Outcome: Count of Participants With Range of Motion (ROM) Full Functional Arc
Description: Range of motion defined as the participant having a full functional arc "Yes" or "No" at 6 month and 12 month post-operative visits.
Time Frame: 6 months and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Number analyzed (Participants) | 106
Participants
  BIORAPTOR™ Knotless Suture Anchor: 6 months: number analyzed (Participants) | 28
  BIORAPTOR™ Knotless Suture Anchor: 6 months: Has full functional arc: Yes | 18
  BIORAPTOR™ Knotless Suture Anchor: 6 months: Has full functional arc: No | 10
  BIORAPTOR™ Knotless Suture Anchor: 6 months: Has full functional arc: Unknown | 0
  BIORAPTOR™ Knotless Suture Anchor: 12 months: number analyzed (Participants) | 15
  BIORAPTOR™ Knotless Suture Anchor: 12 months: Has full functional arc: Yes | 8
  BIORAPTOR™ Knotless Suture Anchor: 12 months: Has full functional arc: No | 7
  BIORAPTOR™ Knotless Suture Anchor: 12 months: Has full functional arc: Unknown | 0
  SpeedLock Hip Suture Anchor: 6 months: number analyzed (Participants) | 78
  SpeedLock Hip Suture Anchor: 6 months: Has full functional arc: Yes | 47
  SpeedLock Hip Suture Anchor: 6 months: Has full functional arc: No | 14
  SpeedLock Hip Suture Anchor: 6 months: Has full functional arc: Unknown | 17
  SpeedLock Hip Suture Anchor: 12 months: number analyzed (Participants) | 18
  SpeedLock Hip Suture Anchor: 12 months: Has full functional arc: Yes | 4
  SpeedLock Hip Suture Anchor: 12 months: Has full functional arc: No | 4
  SpeedLock Hip Suture Anchor: 12 months: Has full functional arc: Unknown | 10

5. Secondary Outcome: Range of Motion (ROM)
Description: Forward flexion angle, internal rotation angle, and external rotation angle captured in degrees based on the physician's Standard of Care.
Time Frame: 6 and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Polyetheretherketone (PEEK) Hip Suture Anchors
Number analyzed (Participants) | 22
degrees
  BIORAPTOR™ Knotless Suture Anchor: Forward Flexion Angle (6 months): number analyzed (Participants) | 10
  BIORAPTOR™ Knotless Suture Anchor: Forward Flexion Angle (6 months) | 97.5 (6.3)
  BIORAPTOR™ Knotless Suture Anchor: Internal Rotation Angle (6 months): number analyzed (Participants) | 2
  BIORAPTOR™ Knotless Suture Anchor: Internal Rotation Angle (6 months) | 10.0 (0)
  BIORAPTOR™ Knotless Suture Anchor: External Rotation (6 months): number analyzed (Participants) | 2
  BIORAPTOR™ Knotless Suture Anchor: External Rotation (6 months) | 37.5 (10.6)
  BIORAPTOR™ Knotless Suture Anchor: Forward Flexion Angle (12 months): number analyzed (Participants) | 7
  BIORAPTOR™ Knotless Suture Anchor: Forward Flexion Angle (12 months) | 102.9 (12.5)
  BIORAPTOR™ Knotless Suture Anchor: Internal Rotation Angle (12 months): number analyzed (Participants) | 2
  BIORAPTOR™ Knotless Suture Anchor: Internal Rotation Angle (12 months) | 35.0 (7.1)
  BIORAPTOR™ Knotless Suture Anchor: External Rotation (12 months): number analyzed (Participants) | 2
  BIORAPTOR™ Knotless Suture Anchor: External Rotation (12 months) | 40.0 (0)
  SpeedLock Hip Suture Anchor: Forward Flexion Angle (6 months): number analyzed (Participants) | 12
  SpeedLock Hip Suture Anchor: Forward Flexion Angle (6 months) | 102.9 (31.8)
  SpeedLock Hip Suture Anchor: Internal Rotation Angle (6 months): number analyzed (Participants) | 2
  SpeedLock Hip Suture Anchor: Internal Rotation Angle (6 months) | 27.5 (24.7)
  SpeedLock Hip Suture Anchor: External Rotation (6 months): number analyzed (Participants) | 2
  SpeedLock Hip Suture Anchor: External Rotation (6 months) | 35.0 (14.1)
  SpeedLock Hip Suture Anchor: Forward Flexion Angle (12 months): number analyzed (Participants) | 4
  SpeedLock Hip Suture Anchor: Forward Flexion Angle (12 months) | 112.8 (11.7)
  SpeedLock Hip Suture Anchor: Internal Rotation Angle (12 months): number analyzed (Participants) | 2
  SpeedLock Hip Suture Anchor: Internal Rotation Angle (12 months) | 16.0 (8.5)
  SpeedLock Hip Suture Anchor: External Rotation (12 months): number analyzed (Participants) | 2
  SpeedLock Hip Suture Anchor: External Rotation (12 months) | 38.5 (9.2)

ADVERSE EVENTS:
Time Frame: Surgery to End of Study (EOS) visit, approximately 12 months
Description: AE reporting was collected retrospectively from the information available in the participant's medical records. A total of 149 participants were enrolled in the study. However, there were 2 participants with multiple devices implanted. Participant Suture Anchor data analyzed independently based on device implanted (i.e., participants implanted with multiple devices were analyzed individually based on unique suture anchor).
Groups:
- BIORAPTOR™ Knotless Suture Anchor: Participants who have received PEEK Suture Anchors in the hip:
  BIORAPTOR™ Knotless Suture Anchor
- SpeedLock Hip Suture Anchor: Participants who have received PEEK Suture Anchors in the hip: SpeedLock Hip Suture Anchor
Arm/Group | BIORAPTOR™ Knotless Suture Anchor | SpeedLock Hip Suture Anchor
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/93
Serious Adverse Events (participants affected / at risk) | 5/58 | 6/93
Other Adverse Events (participants affected / at risk) | 1/58 | 11/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIORAPTOR™ Knotless Suture Anchor (N=58) | SpeedLock Hip Suture Anchor (N=93)
STROKE (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Unrelated to device
POST SURGICAL RIGHT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unlikely related to device
REPEAT LEFT HIP LABRAL TEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unlikely related to device
RIGHT PSOAS TENDONITIS/SNAP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to device
LEFT HIP LABRAL ACETABULAR RETEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated to device
LEFT HIP LABRAL RETEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unlikely related to device
RIGHT HIP LABRAL TEAR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unlikely related to device
LEFT HIP INTRA-ARTICULAR PAIN (General disorders) | 0 (0) | 1 (1) — Unrelated to device
HIP LABRAL TEAR (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Unrelated to device
LEFT HIP LABRAL RETEAR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIORAPTOR™ Knotless Suture Anchor (N=58) | SpeedLock Hip Suture Anchor (N=93)
ILIOPSOAS TENDENOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) — Unrelated to device
RIGHT LEG PAIN (General disorders) | 1 (1) | 0 (0) — Unrelated to device
HIP PAIN (General disorders) | 0 (0) | 4 (4) — Unrelated to device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT03814044/Prot_SAP_000.pdf